CLINICAL TRIAL: NCT02081287
Title: Inositol Hexaphosphate: A Novel Treatment Strategy for Bipolar Disorder?
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: San Diego Veterans Healthcare System (U.S. Federal Agency)
Collaborators: The Depressive and Bipolar Disorder Alternative Treatment Foundation (Other)
Responsible Party: Principal Investigator, Michael McCarthy, Staff Psychiatrist, San Diego Veterans Healthcare System
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DBDAT-2013-MJM
Record Dates: First submitted 2014-03-05; First posted 2014-03-07 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Bipolar Disorder; Manic Depression
Keywords: Bipolar Disorder; Depression; Inositol; Inositol Hexaphosphate; Phytic Acid; IP6; Lithium; Lamotrigine
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — Phytic Acid; Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lamotrigine (Active Comparator): As adjunct to lithium therapy
  Interventions: Drug: Lamotrigine
- IP6 (Experimental): As adjunct to lithium therapy
  Interventions: Drug: IP6

INTERVENTIONS:
Drug: IP6 — IP6 2,000 -3,000 mg per day given orally in two doses
  Other Names: Inositol Hexaphosphate; Phytic Acid
  Arms: IP6
Drug: Lamotrigine — Dose up to 200 mg per day over 10 weeks
  Other Names: Lamictal
  Arms: Lamotrigine

SUMMARY:
Inositol hexaphosphate (IP6, also called inositol hexakisphosphate, and phytic acid) is a naturally occurring phosphorylated derivative of myo-inositol. Myo-inositol has shown preliminary evidence of efficacy in controlling mood symptoms, and good tolerability in bipolar disorder in some studies, but failed to establish efficacy in subsequent meta-analyses. In the investigators proposed work, the investigators plan to orally administer the calcium/magnesium salt of IP6 (2,000-3,000 mg daily in two divided doses) to paid research subjects with a diagnosis of bipolar disorder who are in a depressed state, and who have failed an adequate course of treatment with lithium monotherapy. The investigators hypothesis is that IP6 may be similar to myo-inositol in terms of relieving depression, but more potent and effective. Our aim is conduct a preliminary pilot study in 30 subjects (15 treated with IP6, 15 treated with lamotrigine, an active comparator) to assess the efficacy and tolerability of IP6 as an adjunctive treatment to lithium, the mood stabilizer most commonly used to treat bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

* must have bipolar disorder
* must be currently depressed
* must have failed adequate trial of lithium monotherapy
* must have shown partial response of depression to lithium

Exclusion Criteria:

* diagnoses of schizophrenia, major depression, or other psychotic disorder
* currently pregnant
* unstable medical condition
* active drug or alcohol dependence
* concurrent use of antidepressant or mood stabilizer other than lithium
* active suicidal or homicidal ideation
* past adverse reaction to lamotrigine or current skin rash (lamotrigine arm only)
* history of dietary malabsorption or nutritional deficiency (IP6 arm only)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-05; Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Depression | 10 weeks
  As measured by rater administered Hamilton depression inventory, and Beck Depression Inventory

SECONDARY OUTCOMES:
Sleep Quality | 10 weeks
  As measured by the Pittsburgh Sleep Quality Index
Global Function | 10 weeks
  As measured by the Clinician Global Inventory
Side Effect Burden | 10 weeks
  As measured by standardized inventory
Mania | 10 weeks
  As measured by the Young Mania Scale, and Internal State Scale

OTHER OUTCOMES:
Morning vs Evening Preference | 10 weeks
  As measured by the Basic language morningness scale

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. McCarthy, MD, PhD, Principal Investigator — VA San Diego Healthcare, UCSD
Locations (1):
- VA San Diego Healthcare System, San Diego, California, United States